CLINICAL TRIAL: NCT00618046
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalency Study of Oxcarbazepine 600 mg Tablets Under Fed Conditions
Brief Title: Bioequivalency Study of Oxcarbazepine 600 mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OXCA-T600-PVFD-2
Record Dates: First submitted 2008-01-31; First posted 2008-02-18 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Seizures; Epilepsy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oxcarbazepine

SUMMARY:
The objective of this study was to assess bioequivalence of a potential generic 600 mb oxcarbazepine tablet formulation compared with Novartis Pharmaceutical's 600 mg oxcarbazepine tablet, Trileptal, following a single 600 mg dose, administered with food.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on the physical examination, medical history, or clinical laboratory results at screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with any known enzyme altering drugs.
* History of allergic or adverse response to oxcarbazepine or any other comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2004-11; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two Period, Seven day washout

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Morrison, D.O., Principal Investigator — Bio-Kinetic Clinical Applications, Inc.
Locations (1):
- Bio-Kinetics Clinical Applications, Inc ., Springfield, Missouri, United States